CLINICAL TRIAL: NCT00349349
Title: A Single-arm, International, Multi-center Trial of HuMax-CD20, a Fully Human Monoclonal Anti-CD20 Antibody, in Patients With B-cell Chronic Lymphocytic Leukemia Who Have Failed Fludarabine and Alemtuzumab
Brief Title: HuMax-CD20 in B-Cell Chronic Lymphocytic Leukemia (B-CLL) Patients Failing Fludarabine and Alemtuzumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111773; Hx-CD20-406 (Other: Genmab)
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Leukaemia, Lymphocytic, Chronic
MeSH Terms: conditions — Leukemia, B-Cell | interventions — ofatumumab

ARMS (1):
- ofatumumab (Experimental): Anti-CD20 antibody therapy
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ofatumumab — Intravenous infusion

SUMMARY:
The purpose of this study is to determine whether HuMax-CD20 (ofatumumab) is effective in the treatment of patients failing both fludarabine and alemtuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor cell phenotype consistent with B-CLL
2. Patients with active B-CLL and with an indication for treatment
3. Failing at least one fludarabine-containing treatment regimen
4. Failing at least one alemtuzumab-containing treatment regimen
5. ECOG Performance Status of 0, 1, or 2
6. Life expectancy of at least 4 months

Exclusion Criteria:

1. Previous treatment with alemtuzumab within 6 weeks prior to Visit 2
2. Previous autologous stem cell transplantation within 6 months prior to Visit 2
3. Allogeneic stem cell transplantation
4. Radioimmunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Wierda WG, Padmanabhan S, Chan GW, Gupta IV, Lisby S, Osterborg A; Hx-CD20-406 Study Investigators. Ofatumumab is active in patients with fludarabine-refractory CLL irrespective of prior rituximab: results from the phase 2 international study. Blood. 2011 Nov 10;118(19):5126-9. doi: 10.1182/blood-2011-04-348656. Epub 2011 Aug 19. PMID 21856867
- [Result] Wierda WG, Kipps TJ, Mayer J, Stilgenbauer S, Williams CD, Hellmann A, Robak T, Furman RR, Hillmen P, Trneny M, Dyer MJ, Padmanabhan S, Piotrowska M, Kozak T, Chan G, Davis R, Losic N, Wilms J, Russell CA, Osterborg A; Hx-CD20-406 Study Investigators. Ofatumumab as single-agent CD20 immunotherapy in fludarabine-refractory chronic lymphocytic leukemia. J Clin Oncol. 2010 Apr 1;28(10):1749-55. doi: 10.1200/JCO.2009.25.3187. Epub 2010 Mar 1. PMID 20194866
- [Derived] Struemper H, Sale M, Patel BR, Ostergaard M, Osterborg A, Wierda WG, Hagenbeek A, Coiffier B, Jewell RC. Population pharmacokinetics of ofatumumab in patients with chronic lymphocytic leukemia, follicular lymphoma, and rheumatoid arthritis. J Clin Pharmacol. 2014 Jul;54(7):818-27. doi: 10.1002/jcph.268. Epub 2014 Jan 28. PMID 24443277

RESULTS

PARTICIPANT FLOW:
Groups:
- 2000 mg Ofatumumab + DR: Ofatumumab intravenous (iv) infusion was initiated at 300 milligrams (mg), followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The independent endpoint review committee (IRC) classified these participants as double refractory (DR), defined as participants who were enrolled in the study and were refractory to both fludarabine and alemtuzumab.
- 2000 mg Ofatumumab + BFR: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The IRC classified these participants as bulky fludarabine refractory (BFR), defined as participants who were enrolled in the study and were refractory to fludarabine with bulky lymphadenopathy.
- 2000 mg Ofatumumab + Other: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The IRC classified these participants as "other," defined as participants who were enrolled in the study but did not meet criteria for DR or BFR.
Period: Overall Study
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Started | 95 | 112 | 16
Completed | 42 | 50 | 10
Not Completed | 53 | 62 | 6
Not completed — Adverse Event | 5 | 6 | 2
Not completed — Withdrawal by Subject | 5 | 2 | 1
Not completed — Withdrawn due to Disease Progression | 27 | 37 | 1
Not completed — Death | 13 | 10 | 1
Not completed — Other Treatment Selected | 2 | 0 | 0
Not completed — Participant Reduced General Condition | 0 | 1 | 0
Not completed — Physician Decision | 1 | 2 | 1
Not completed — No Response | 0 | 3 | 0
Not completed — New Malignancy (Bladder Cancer) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2000 mg Ofatumumab + DR: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The IRC classified these participants as DR, defined as participants who were enrolled in the study and were refractory to both fludarabine and alemtuzumab.
- 2000 mg Ofatumumab + BFR: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The IRC classified these participants as BFR, defined as participants who were enrolled in the study and were refractory to fludarabine with bulky lymphadenopathy.
- 2000 mg Ofatumumab + Other: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. The IRC classified these participants as "other,"defined as participants who were enrolled in the study but did not meet criteria for DR or BFR.
- Total: Total of all reporting groups
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other | Total
Number analyzed (Participants) | 95 | 112 | 16 | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.4) | 64.4 (9.3) | 64.5 (7.4) | 63.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 31 | 5 | 60
  Male | 71 | 81 | 11 | 163
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1 | 2
  Black or African American | 2 | 1 | 0 | 3
  Hispanic or Latino | 1 | 0 | 0 | 1
  White | 88 | 111 | 15 | 214
  Arab | 1 | 0 | 0 | 1
  Yemenite | 1 | 0 | 0 | 1
  Middle Eastern | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) Classified as Responders and Non-responders for Objective Response as Assessed by an Independent Endpoint Review Committee (IRC) in Accordance With the National Cancer Institute Working Group (NCIWG) 1996 Guidelines
Description: Par. with complete remission (CR), nodular partial remission (nPR), and partial remission (PR) were classified as responders, while those with stable disease (SD) and progressive disease (PD) were classified as non-responders. Per the NCIWG guideline (1996): CR; no lymphadenopathy/hepatomegaly/splenomegaly/constitutional symptoms, normal hematology, bone marrow sample as normocellular for age, <30% lymphocytes (LC), no lymphoid nodule; PR: a >=50% decrease in LC/lymphadenopathy; nPR: persistent nodules in bone marrow; PD: new lesion or increase by >=50% from baseline; SD: no CR, PR, or PD.
Time Frame: Start of treatment (Week 0 of Visit 2) until Week 24
Population: Full Analysis Set (FAS): all participants who had been exposed to study drug irrespective of their compliance to the planned course of treatment. Participants not evaluable (NE) were due to patient withdraw, refusal, non-trial drug related AEs, and death
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
participants
  Responders with CR | 0 | 2 | 0
  Responders with nPR | 0 | 0 | 1
  Responders with PR | 47 | 46 | 9
  Non-responders with SD | 33 | 52 | 4
  Non-responders with PD | 5 | 9 | 1
  NE | 10 | 3 | 1
Statistical Analysis 1: Comparison: 2000 mg Ofatumumab + DR; Test type: Superiority or Other; p < 0.0001, Two-sided exact binomial test — The p value is testing the hypothesis that the response rate is equal to 15% versus the response rate is not equal to 15%; percentage of responders = 0.49, 95.3% CI 2-sided [0.39 to 0.60] — Two-sided 95.3% exact confidence intervals were calculated based on the binomial distribution
Statistical Analysis 2: Comparison: 2000 mg Ofatumumab + BFR; Test type: Superiority or Other; p < 0.0001, Two-sided exact binomial test — [p-value comment as in outcome 1, analysis 1]; percentage of responders = 0.43, 95.3% CI 2-sided [0.33 to 0.53] — Two sided 95.3% exact confidence intervals were calculated based on the binomial distribution
Statistical Analysis 3: Comparison: 2000 mg Ofatumumab + Other; Test type: Superiority or Other; p < 0.001, Two-sided exact binomial test — [p-value comment as in outcome 1, analysis 1]; percentage of responders = 0.63, 95.3% CI 2-sided [0.35 to 0.85] — Two-sided 95.3% exact confidence intervals were calculated based on the binomial distribution

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the initial response (first visit at which response is observed) to progression or death. If the participant had progression between scheduled visits, no progression at the end of the trial, treatment discontinuation for undocumented progression, treatment discontinuation for toxicity or other reason, new anti-cancer treatment, and experienced death or progression after two or more missed visits in a row the endpoint was censored.
Time Frame: Start of treatment (Week 0 of Visit 2) until Week 24
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
months | 5.5 [3.7 to 7.2] | 6.4 [4.6 to 7.0] | 7.4 [2.8 to 12.4]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization until progression/death. Per the IRC, if the participant had progression between scheduled visits, died before the first assessment, or died between adequate visits, the endpoint was considered progressed. If there was no progression at the end of the trial, treatment discontinuation for undocumented progression, treatment discontinuation for toxicity/other reason, new anti-cancer treatment, and death/progression after 2 or more missed visits in a row, the endpoint was censored. Clinical progression is not considered as progression endpoint.
Time Frame: Start of treatment (Week 0 of Visit 2) until Week 24
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
months | 4.6 [3.9 to 6.3] | 5.5 [4.6 to 6.4] | 8.9 [3.7 to 11.8]

4. Secondary Outcome: Time to Next Chronic Lymphocytic Leukemia (CLL) Treatment
Description: Time to next chronic lymphocytic leukemia (CLL) treatment is defined as the time from treatment allocation/randomization (Visit 2) until the time of the first administration of the next CLL treatment other than ofatumumab (or HuMaxCD20, a fully human monoclonal antibody to CD20 that is expressed on the surface of B-cells).
Time Frame: Time from randomization (Week 0 of Visit 2) until the time of first administration of a CLL treatment other than ofatumumab (assessed for a median of 8.7 weeks currently [or up to 13.3 months])
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
months | 8.5 [7.2 to 9.9] | 8.2 [7.0 to 9.3] | 12.1 [8.2 to 14.7]

5. Secondary Outcome: Overall Survival
Description: OS is defined as the time from allocation to death. OS will also be subgrouped for responders and non-responders.
Time Frame: Start of randomization (Week 0 of Visit 2) until death (up to a median of 17.1 weeks)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
months | 13.9 [9.8 to 18.6] | 17.4 [15.0 to 24.5] | 28.3 [19.0 to 29.2]

6. Secondary Outcome: Percent Change From Baseline to Week 7 in Peripheral CD5+CD19+ Cell Counts
Description: The peripheral blood for each participant was collected and analyzed for CD5+CD19+ cell counts. CD is "cluster of differentiation," is a cell surface marker for immunophenotyping, and, in this case, is a surrogate for B cell malignancy (indicates malignant B cells). Percent change from Visit 2 (Week 0, Baseline) = (value at Week 7 minus value at Week 0 divided by value at Week 0) x 100.
Time Frame: Baseline (Visit 2) until Week 7 (Visit 9)
Population: FAS
Measure: Median (Full Range); unit: percent change in cell counts
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
percent change in cell counts | -93 [-100 to 597] | -92 [-100 to 1384] | -95 [-100 to 640]

7. Secondary Outcome: Percent Change From Baseline to Week 7 in Peripheral CD5+CD20+ Cell Counts
Description: The peripheral blood for each participant was collected and analyzed for CD5+CD20+ cell counts. CD is "cluster of differentiation," is a cell surface marker for immunophenotyping, and, in this case, is a surrogate for B cell malignancy (indicates malignant B cells). Percent change from Visit 2 (Week 0, Baseline) = (value at Week 7 minus value at Week 0 divided by value at Week 0) x 100.
Time Frame: Baseline (Visit 2) until Week 7 (Visit 9)
Population: FAS
Measure: Median (Full Range); unit: percent change in cell counts
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
percent change in cell counts | -100 [-100 to 236] | -100 [-100 to -13] | -100 [-100 to -96]

8. Secondary Outcome: Median Percent Change of Tumor Size (Sum of Products Dimensions [SPD]) From Baseline (Visit 2) to Week 24 (Visit 14)
Description: Tumor size and change in tumor size will be measured by the absolute value of and the percent change in the sum of products of the diameters of the largest abnormal lymph nodes from Baseline to Week 24 (Visit 14). Percent change from Visit 2 (Baseline, Week 0) = (value at Week 24 minus value at Week 0 divided by value at Week 0) x 100.
Time Frame: Baseline (Visit 2) until Week 24 (Visit 14)
Population: FAS
Measure: Median (Full Range); unit: percent change in tumor size
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
percent change in tumor size | -81 [-100 to 100] | -80 [-100 to 335] | -82 [-100 to -6]

9. Secondary Outcome: Number of Participants With Complete Resolution of Constitutional Symptoms at Week 24
Description: Participants with complete resolution of constitutional symptoms were those in whom no constitutional symptoms, such as night sweats, weight loss, and fever or extreme fatigue, were observed.
Time Frame: Baseline (Visit 2) and Week 24
Population: FAS. Data were provided for the number of participants with constitutional symptoms at baseline attending each visit. Participants withdrawn during the study were not analyzed. (Participants without baseline constitutional symptoms did not experience new constitutional symptoms during the trial period.)
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 42 | 57 | 10
participants | 34 | 46 | 9

10. Secondary Outcome: Number of Participants With Complete Resolution of Lymphadenopathy
Description: Participants with complete resolution of lymphadenopathy (disease involving the lymph nodes) were defined as those in whom all observed lymph nodes were of normal size (all nodes <1 centimeters) as determined by physical examination assessed by the investigator. All palpable lymph node sizes were recorded.
Time Frame: Baseline (Visit 2) to end of study (up to Week 24)
Population: FAS. Data were provided for the number of participants with lymphadenopathy at baseline attending each visit. Participants withdrawn during the study were not analyzed. (Participants without baseline lymphadenopathy remained free of lymphadenopathy during the trial.)
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 82 | 100 | 13
participants | 27 | 18 | 6

11. Secondary Outcome: Number of Participants With Improvement on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale at Week 24
Description: ECOG performance status is a measure of the participant's ability to carry out activities of daily living on 6-point scale (0=fully active, 1=restricted in physically activity, ambulatory, 2=ambulatory [>50% of waking hours], 3=capable of only limited self care, 4=completely disabled, 5=Dead). Improvement in ECOG performance status is defined as a decrease from baseline by at least one score on the ECOG scale.
Time Frame: Baseline (Visit 2) and Week 24
Population: FAS. Data were provided for participants (par.) with an ECOG score >0 at baseline attending each visit. Par. withdrawn from the study were not analyzed. (55 par. had an ECOG performance status of 0 at baseline and therefore did not have the opportunity to improve. No par. with an ECOG score of 0 at baseline worsened during the trial.)
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 55 | 70 | 12
participants | 25 | 35 | 7

12. Secondary Outcome: Number of Participants Who Were Positive, Negative, or Had Missing Data for the Indicated Fluorescence in Situ Hybridization (FISH) Prognostic Factors at Screening
Description: The number of participants (par.) who were positive, negative, or had missing data for the following prognostic factors indicative of altered responsiveness to treatment and/or survival was measured: 17p-, 11q-, +12q, 6q-, 13q-. Par. were assessed by FISH for these chromosomal abnormalities known tobe prognostic for time to treatment and survival when detected at diagnosis. Par. were categorized by the chromosomal abnormality detected: 17 p deletion, 11q deletion (but not 17 p deletion), 12 q trisomy (but not 17 p or 111q deletion), 13q deletion only, and no chromosomal abnormalities found.
Time Frame: Screening (Visit 1, <=14 days prior to Visit 2)
Population: FAS. Par. were categorized hierarchically (by severity of abnormality): par. with a 17 p deletion (D); par. with an 11q D, but not a 17 p D; par. with 12q trisomy, but not a 17p or 11q D; par. with no aberrations found; par. with a 13q D as the sole aberration; and par. with 6q D (and not any of the above categories). Some par. had missing data.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 92 | 110 | 16
participants
  FISH 17p-, negative | 64 | 89 | 14
  FISH 17p-, positive | 27 | 19 | 1
  FISH 17p-, missing | 4 | 4 | 1
  FISH 11q-, negative | 56 | 69 | 11
  FISH 11q-, positive | 36 | 41 | 5
  FISH 11q-, missing | 3 | 2 | 0
  FISH +12q, negative | 76 | 91 | 11
  FISH +12q, positive | 15 | 19 | 5
  FISH +12q, missing | 4 | 2 | 0
  FISH 6q-, negative | 89 | 101 | 15
  FISH 6q-, positive | 2 | 9 | 0
  FISH 6q-, missing | 4 | 2 | 1
  FISH 13q-, negative | 46 | 53 | 9
  FISH 13q-, positive | 45 | 57 | 7
  FISH 13q-, missing | 4 | 2 | 0

13. Secondary Outcome: Number of Participants With Improvement in Hemoglobin
Description: The number of participants (par.) who had improvement in hemoglobin levels >=11 grams (g)/deciliter (dl) (6.8 millimoles/liter) or 50% improvement over baseline was measured.
Time Frame: Baseline (Visit 2) to Week 28
Population: FAS. Par. were excluded from analysis if they received treatment of red blood cells (RBCs), received transfusions or a RBC growth factor (erythropoietin), died, withdrew from the trial, or began next CLL treatment. Only those par. remaining in the study at Week 28 were analyzed. No par. in the "Other" treatment arm met the criteria for analysis.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 49 | 62 | 8
participants | 18 | 20 | 5

14. Secondary Outcome: Number of Participants With Improvement in Thrombocytopenia (Thromb.)
Description: Improvement in thromb. is defined as a decrease from Visit 2 by >=1 National Cancer Institute Common Terminology Criteria (NCI CTC) grade. Thromb. is defined as low platelet counts resulting from refractory CLL, damage from prior treatment, advanced age, or reduced bone marrow function and can be considered as an adverse condition. Adverse events (AEs) such as thromb. in a cancer indication are graded on a scale determined by the NCI called the NCI CTC: lowest, grade 1; highest, grade 5 (death). Changes in this grading can assess improvements or declines in the severity of the AE.
Time Frame: Baseline (Visit 2) to Week 28
Population: FAS. Only those participants remaining in the study at Week 28 were analyzed. No par. in the "Other" treatment arm met the criteria for analysis.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 10 | 13 | 0
participants | 4 | 6 |

15. Secondary Outcome: Number of Participants With Complete Resolution of Hepatomegaly
Description: Participants with complete resolution of enlarged liver (hepatomegaly) were defined as those with an enlarged palpable liver at baseline followed by the absence of hepatomegaly post- baseline (i.e., the liver was of normal size). Liver size was assessed by physical examination and documented as "centimeters" under the costal margin with relative changes in spleen size in 1 dimension calculated based on palpated numeric measurements (as per the 1996 NCIWG guidelines).
Time Frame: Baseline (Visit 2) until Week 24
Population: FAS. Data were provided for the number of participants with hepatomegaly from baseline attending each visit. Participants withdrawn during the study were not analyzed. Only participants with baseline hepatomegaly and a post-baseline assessment are included.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 21 | 28 | 7
participants | 17 | 19 | 4

16. Secondary Outcome: Number of Participants With Improvement in Neutropenia
Description: Low levels of neutrophils (neutropenia) may increase the risk of developing serious infections and may be considered an adverse condition and evaluated on the NCI CTC with a grade. Improvement in neutropenia is defined as a decrease from Visit 2 (baseline) by at least one NCI CTC grade. Improvement is defined as a decrease from Visit 2 by at least one NCI CTC grade.
Time Frame: Baseline (Visit 2) to Week 28
Population: FAS. Only those par. remaining in the study at Week 28 were analyzed. No par. in the "Other" treatment arm met the criteria for analysis.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 30 | 25 | 3
participants | 20 | 17 | 1

17. Secondary Outcome: Number of Participants With Complete Resolution of Splenomegaly
Description: Participants with complete resolution of enlarged spleen (splenomegaly) were defined as those with an enlarged palpable spleen at baseline followed by the absence of splenomegaly post-baseline (i.e., the spleen was of normal size). Spleen size was assessed by physical examination and documented as "centimeters" under the costal margin with relative changes in spleen size in 1 dimension calculated based on palpated numeric measurements (as per the 1996 NCIWG guidelines).
Time Frame: Baseline (Visit 2) until Week 24
Population: FAS. Data were provided for the number of participants with splenomegaly at baseline attending each visit. Participants withdrawn during the study were not analyzed. Only participants with baseline splenomegaly and a post-baseline assessment are included.
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 43 | 63 | 10
participants | 28 | 38 | 5

18. Secondary Outcome: Number of Participants Who Experienced Any Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. A list of AEs experienced in the study with a frequency threshold of 5% can be found in the AE section of this results record.
Time Frame: From first infusion (Visit 2/Week 0) to Visit 21 (Month 24 of follow-up [up to Month 48]) or time of withdrawal (treatment and follow-up)
Population: FAS
Measure: Number; unit: participants
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Number analyzed (Participants) | 95 | 112 | 16
participants | 90 | 107 | 16

19. Secondary Outcome: Cmax and Ctrough at Dose 1 (Visit 2, Week 0), Dose 8 (Visit 9, Week 7), and Dose 12 (Visit 14, Week 24)
Description: Cmax is defined as the maximum concentration of drug in serum samples. Ctrough is defined as the trough serum concentration (measured concentration at the end of a dosing interval [taken directly before the next administration]). No drug was present before the first infusion; therefore, there are no Ctrough results for Dose 1
Time Frame: Visit 2 (Week 0), Visit 9 (Week 7), and Visit 14 (Week 24)
Population: FAS. Data were provided for the number of participants attending each visit. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams per liter (mg/L)
Groups:
- 2000 mg Ofatumumab + Total: Ofatumumab iv infusion was initiated at 300 mg, followed by seven weekly 2000 mg infusions and then four monthly infusions of 2000 mg for a duration of 24 weeks. Data from all three groups of participants (DR, BFR, and Other) have been combined.
Arm/Group | 2000 mg Ofatumumab + Total
Number analyzed (Participants) | 215
Milligrams per liter (mg/L)
  Cmax at Dose 1, n=215 | 61.4 (0.73)
  Ctrough at Dose 8, n=192 | 549 (2.34)
  Cmax at Dose 8, n=193 | 1391 (0.46)
  Ctrough at Dose 12, n=106 | 32.1 (58.8)
  Cmax at Dose 12, n=106 | 827 (0.41)

20. Secondary Outcome: AUC (0-inf) and AUC(0-tau) at Dose 8 (Visit 9, Week 7) and Dose 12 (Visit 14, Week 24)
Description: AUC is defined as the area under the ofatumumab concentration-time curve as a measure of drug exposure. AUC(0-inf) is AUC from the start of infusion extrapolated to infinity. AUC(0-tau) is AUC from the start of infusion over the dosing interval.
Time Frame: Visit 9 (Week 7) and Visit 14 (Week 24)
Population: FAS. Data were provided for the number of participants attending each visit for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams x hour per liter (mg.h/L)
Arm/Group | 2000 mg Ofatumumab + Total
Number analyzed (Participants) | 163
Milligrams x hour per liter (mg.h/L)
  AUC(0-inf) at Dose 8, n=133 | 463418 (0.94)
  AUC(0-inf) at Dose 12, n=83 | 203536 (1.64)
  AUC(0-tau) at Dose 8, n=163 | 171286 (0.48)
  AUC(0-tau) at Dose 12, n=84 | 165617 (1.23)

21. Secondary Outcome: Half-life (t1/2) at Dose 8 (Visit 9, Week 7) and at Dose 12 (Visit 14, Week 24)
Description: Half-life ( t1/2) is defined as the terminal half-life and is the time required for the amount of drug in the body to decrease by half.
Time Frame: Visit 9 (Week 7) and Visit14 (Week 24)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 2000 mg Ofatumumab + Total
Number analyzed (Participants) | 141
hours
  t1/2 at Dose 8, n=141 | 326 (0.56)
  t1/2 at Dose 12, n=81 | 277 (0.87)

22. Secondary Outcome: Clearance (CL) After Dose 8 (Visit 9, Week 7) and Dose 12 (Visit 14, Week 24)
Description: CL is the clearance of drug from serum, which is defined as the volume of serum from which the drug is cleared per unit time.
Time Frame: Visit 9 (Week 7) and Visit 14 (Week 24)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per hour (mL/h)
Arm/Group | 2000 mg Ofatumumab + Total
Number analyzed (Participants) | 163
Milliliters per hour (mL/h)
  CL at Dose 8, n=163 | 11.7 (0.48)
  CL at Dose 12, n=84 | 12.1 (1.23)

23. Secondary Outcome: Volume of Distribution at Steady State (Vss) at Dose 8 (Visit 9, Week 7) and at Dose 12 (Visit 14, Week 24)
Description: Vss is defined as the volume of distribution at steady state of ofatumumab.
Time Frame: Visit 9 (Week 7) and Visit 14 (Week 24)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | 2000 mg Ofatumumab + Total
Number analyzed (Participants) | 133
Liters (L)
  Vss at Dose 8, n=133 | 4.84 (0.30)
  Vss at Dose 12, n=83 | 3.73 (0.30)

ADVERSE EVENTS:
Arm/Group | 2000 mg Ofatumumab + DR | 2000 mg Ofatumumab + BFR | 2000 mg Ofatumumab + Other
Serious Adverse Events (participants affected / at risk) | 60/95 | 59/112 | 12/16
Other Adverse Events (participants affected / at risk) | 90/95 | 107/112 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2000 mg Ofatumumab + DR (N=95) | 2000 mg Ofatumumab + BFR (N=112) | 2000 mg Ofatumumab + Other (N=16)
Pneumonia (Infections and infestations) | 12 | 12 | 2
Sepsis (Infections and infestations) | 5 | 6 | 0
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 4 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 3 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Aspergilloma (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Enterocolitis infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fusarium infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Injection site infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Progessive multifocal (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Hemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Anemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytic infiltration (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Disease progression (General disorders) | 4 | 5 | 1
Pyrexia (General disorders) | 6 | 4 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 0
Cardic failure (Cardiac disorders) | 1 | 1 | 0
Myopericarditis (Cardiac disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Chronic lympocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Hodgkins disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lower respiration infection (Infections and infestations) | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Enterocolitis infections (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Eye infection staphylococcal (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 1 | 0
Pseuromonas infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 0
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute repiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cerebral ischemia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Immunodeficiency (Immune system disorders) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Pyroderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2000 mg Ofatumumab + DR (N=95) | 2000 mg Ofatumumab + BFR (N=112) | 2000 mg Ofatumumab + Other (N=16)
Fatigue (General disorders) | 12 | 22 | 1
Pyrexia (General disorders) | 22 | 18 | 7
Oedema peripheral (General disorders) | 9 | 14 | 1
Chills (General disorders) | 13 | 13 | 2
Pneumonia (Infections and infestations) | 15 | 15 | 4
Bronchitis (Infections and infestations) | 14 | 12 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 17 | 2
Nasopharyngitis (Infections and infestations) | 10 | 10 | 1
Herpes zoster (Infections and infestations) | 6 | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 24 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12 | 3
Anemia (Blood and lymphatic system disorders) | 17 | 20 | 2
Neutropenia (Blood and lymphatic system disorders) | 19 | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 16 | 16 | 5
Nausea (Gastrointestinal disorders) | 13 | 15 | 1
Rash (Skin and subcutaneous tissue disorders) | 17 | 8 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 9 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 7 | 2
Hypotension (Vascular disorders) | 7 | 6 | 1
Insomnia (Psychiatric disorders) | 7 | 7 | 1
Headache (Nervous system disorders) | 8 | 5 | 1
Sinusitis (Infections and infestations) | 7 | 7 | 1
Urinary tract infection (Infections and infestations) | 4 | 8 | 1
Lower respiratory tract infections (Infections and infestations) | 5 | 6 | 3
Vomiting (Gastrointestinal disorders) | 7 | 7 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4 | 0
Parasthesia (Nervous system disorders) | 5 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.